CLINICAL TRIAL: NCT05512195
Title: Safety and Efficacy of a New Approach to Delineating Clinical Target Volume by Referencing the Nerve Fiber Bundles for Radiotherapy of Glioblastoma
Brief Title: Safety and Efficacy of a New Approach to Delineating Clinical Target Volume of Glioblastoma
Acronym: GBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhongnanH GBM
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Glioblastoma
Keywords: Radiotherapy, clinical target volume, Glioblastoma multiforme (GBM), radiation volume, the white matter tracts.
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New delineation approach （NDA）group (Experimental): use a new method for clinical target volume delineation by referencing the nerve fiber bundles
  Interventions: Radiation: New delineation approach

INTERVENTIONS:
Radiation: New delineation approach — New delineation approach

SUMMARY:
Radiotherapy (RT) is one of the most important local treatments besides surgery, but currently, no consensus has been made regarding the optimal radiation volume for high grade gliomas. The most main growth characteristics of glioblastoma is infiltrative growth through the white matter tracts, regions along the white matter tracts especially at the direction of the main fiber bundles would have a higher risk of microscopic tumor cell dissemination. However, in current practice, recommends for the CTV definition is adding a 2 cm symmetrical margin to GTV or peritumoral edema in all directions, which hardly account for the growth characteristics of gliomas that are known from histopathological findings.

DETAILED DESCRIPTION:
Patients with glioblastoma were recruited for this study based on the following eligibility criteria: Age between 18 and 70, performance status of 0-1 (Eastern Cooperative Oncology Group performance status), histologically confirmed glioblastoma, no cerebrospinal fluid and distant metastatic disease. All patients had adequate hematologic, hepatic, and renal function. Patients younger than 18 years; patients with a prior (i.e. within 5 years) or synchronous malignancy, other than non-melanoma skin cancer; and those with significant comorbidities were excluded.

Eligible patients received chemoradiotherapy (CRT) ( PTV-GTV: 60Gy at 2.0Gy per fraction, 5 fractions per week for 6 weeks; PTV-CTV: 54Gy at 1.8Gy per fraction, 5 fractions per week for 6 weeks) with a Temozolomide (TMZ) regimen（75mg/m2 per day during RT）, followed by 6 additional cycles of TMZ. (150 mg/m2 for the first cycle and 200 mg/m2 for the 2-6th cycles, on days 1-5, every 4 weeks) .

The investigators established a detailed protocol for target delineation of the CTV based on brain anatomy, white mater fiber tracts distribution and the growth patterns of tumor. Briefly, along the directions of the main nerve fiber bundles ，the CTV is defined as peritumoral edema plus 1cm. while in other directions, the CTV is defined as GTV plus 2cm and should be adjusted to anatomical borders such as the skull (0 mm, using bone window), ventricles (5 mm), falx (0 mm), tentorium cerebelli (0 mm), visual pathway/optic chiasm and brainstem (each 0 mm) and modified to include all regions of abnormal T2/FLAIR MRI signal. Deep brain white matter is the focus for RT target contour, regions of normal uninvolved gray matter should be modified to be protected.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* performance status of 0-1 (Eastern Cooperative Oncology Group performance status)
* histologically confirmed glioblastoma
* no cerebrospinal fluid and distant metastatic disease
* All patients had adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

* younger than 18 years;
* patients with a prior (i.e. within 5 years) or synchronous malignancy, other than non-melanoma skin cancer; and those with significant comorbidities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  Time from the start of treatment to death due to the disease

SECONDARY OUTCOMES:
recurrence-free survival (RFS) | 1 year
  Time from the start of treatment to recurrence

IPD SHARING:
Plan to Share IPD: Undecided